CLINICAL TRIAL: NCT01809080
Title: Investigation Into the Interaction Between Genes and Stress in the Etiology of Depression in Interns
Brief Title: Intern Health Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Srijan Sen, Assistant Professor of Psychiatry, Medicial School, University of Michigan
Other Study IDs: MH-095109
Record Dates: First submitted 2013-03-01; First posted 2013-03-12 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2024-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva: DNA collection kits are sent via postal mail and participants are asked to provide a small sample of saliva.
  Blood samples (up to 50 mL via venopuncture): whole blood and serum will be assessed.
  Hair: The total diameter taken from the scalp's posterior vertex will be about 3 mm, which is about half of the diameter of pencil (approximately 100 hair strands with a minimum of 50 mg of hair for a 3-cm segment).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (20):
- 2020
- 2019
- 2018
- 2017
- 2016
- 2015
- 2014
- 2013
- 2012
- 2011
- 2010
- 2009
- 2008
- 2007
- 2021
- 2022
- 2023
- 2024
- 2025
- 2026

SUMMARY:
Retrospective studies have established a strong correlation between reports of life stress and depression. Investigators have begun to further explore this relationship by examining the role of gene x stress interactions in the pathogenesis of depression. In a recent landmark study, Caspi and colleagues (2003) reported an interaction between a serotonin transporter promoter polymorphism and life stress in the development of depression. This finding has been replicated in some but not all follow up studies. Despite the initial promise of these results, the ability to draw definitive conclusions is compromised by significant study design limitations: 1) retrospective design 2) a focus on acute rather than chronic stress 3) substantial variation in the character and intensity of stress between subjects. Medical internship is a period filled with predictable and high levels of chronic uncontrolled stress. Rates of depression among interns are elevated compared to the general population. In this study, we aim to utilize the predictable and consistent stress of internship to investigate the relationship between stress, genes and depression with a prospective study design that bypasses some of the pitfalls of previous studies.

DETAILED DESCRIPTION:
Specific Aims Retrospective studies have established a strong correlation between reports of life stress and depression. Investigators have begun to further explore this relationship by examining the role of gene x stress interactions in the pathogenesis of depression. In a recent landmark study, Caspi and colleagues (2003) reported an interaction between a serotonin transporter promoter polymorphism and life stress in the development of depression. This finding has been replicated in some but not all follow up studies. Despite the initial promise of these results, the ability to draw definitive conclusions is compromised by significant study design limitations: 1) retrospective design 2) a focus on acute rather than chronic stress 3) substantial variation in the character and intensity of stress between subjects. Medical internship is a period filled with predictable and high levels of chronic uncontrolled stress. Rates of depression among interns are elevated compared to the general population. In this study, we aim to utilize the predictable and consistent stress of internship to investigate the relationship between stress, genes and depression with a prospective study design that bypasses some of the pitfalls of previous studies.

Goal 1) Assess the prevalence and development of depression among medical interns

Although small studies have assessed the point prevalence of depression among medical residents, no study has prospectively followed the development of depressive symptoms through residency. We will collect baseline psychological profiles of incoming interns prior to the commencement of residency duties and subsequently assess for depressive symptoms at 3-month intervals throughout internship. This data will allow us to:

1. Assess the point prevalence of depression among interns in a large sample.
2. Determine the change in depressive symptoms through the course of the intern year
3. Evaluate stable psychological factors that associate with the development of depression in the face of life stress.

Goal 2) Evaluate the presence of genotype x stress interaction among this sample

1. There is conflicting evidence concerning the presence of an interaction between the serotonin transporter promoter polymorphism (5-HTTLPR) and life stress in the development of depression. We will assess the presence and strength of this interaction in the sample of medical interns using a study design that avoids many of the pitfalls affecting previous studies.
2. We will explore novel putative interactions between stress and genetic variants in additional genes including BDNF, CRH, COMT, serotonin 1A and serotonin 2A receptor variants in the development of depression.

Goal 3) Evaluate the relationship between serum endothelial and immune factors and the development of depressive symptoms under stress.

The identification biomarkers that predict the onset of depression can facilitate more timely and accurate identification of individuals at high risk for the disorder. Unfortunately appropriate studies are lacking, largely because it is difficult to know exactly when a depressive episode will occur. Medical internship represents a rare situation where we can prospectively predict when a cohort of individuals shift will shift from a low stress environment to a high stress environment and thus predict when this cohort will experience a dramatic increase in depressive symptoms.

Goal 4) Examine the temporal relationship between hair cortisol levels, stress exposure and development of depressive symptoms.A novel technique allows us to assess chronic HPA axis activity by measuring cortisol in the growing hair, providing an integrated measure of total cortisol secretion over extended periods of time (1-3 months).

By incorporating this novel method into an established longitudinal study of a chronic stressor that dramatically increases rates of depression, we have a unique opportunity to determine a) whether cortisol levels prior to stress exposure predict risk of depression in response to the stressor (b) whether cortisol rise in response to stress exposure precedes and perhaps contributes to development of depressive symptoms or whether cortisol elevations in depression develop after symptom onset and perhaps reflect a consequence of depression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for our study will be drawn from incoming interns in the traditional and primary care internal medicine, general surgery, pediatrics, obstetrics/gynecology, neurology and psychiatry residency programs at participating University and Community residency programs, as well as fourth year medical students at participating medical schools.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical internship is an attractive model to bypass some limitations of previous studies. Internship is well chronicled as a time of high stress (Butterfield 1988; Addison et al 2004). Interns are faced with long work hours, sleep deprivation, loss of autonomy and extreme emotional situations (Shanafelt & Habermann 2002). Many physicians recall internship as among the most stressful years of their lives (Duffy 2005). The stress of internship is often uncontrollable, unpredictable and chronic; features that are particularly linked to the development of depression (Kendler et al 2003; Cryan et al 2004). Several studies have estimated the point prevalence of depression among interns at 28%-37% (Valko & Clayton 1975; Reuben 1985; Cohen et al 2006), in contrast to a point prevalence of 5% in general population (Murphy et al 2000). There is also evidence that physicians have underlying personality traits that predispose to depression (McDonough 1990; Hojat et al 1999).
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2007-05; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assess the change in rates of depression among medical interns. | Months 0, 3, 6, and 12 of Intern Year
  The point prevalence of depression at various points through internship will be determined using subject responses to DSM-IV major depression items at the 0, 3-month, 6-month and 12-month assessments. To investigate whether there is a significant change in depressive symptoms through intern year, the investigators will compare PHQ (baseline) and PHQ (6 month) depression scores through a paired T-test. The effect of baseline psychological traits (neuroticism, resilience, personal history of depression, family history of depression, early family environment, social supports) on the development of depression will also be explored through linear regression analyses with each of the psychological factors as independent variables and PHQ (change) [PHQ (6 month) - PHQ (baseline)] as the dependent variable. The investigators will use linear regression to investigate correlations between training program characteristics (average work hours, specialty) and PHQ (change).

SECONDARY OUTCOMES:
Evaluate the presence of genotype x stress interaction among this sample. | Sample within first 6 months of Intern Year (Because DNA sequence generally does not change with time, the exact timing of sample collection is not critical to the analysis)
  As a baseline analysis, the investigators will investigate association between each variant/haplotype and PHQ (baseline) scores using linear regression. To explore gene x environment interactions, the investigators will assess for association between each variant/haplotype and PHQ change scores (Mean (3,6,9 and 12 month PHQ score) - Baseline (PHQ score)).
Evaluate the relationship between serum factors and changes in depressive symptoms under stress. | Months 0 and 10 of Intern Year
  For each of the proteins assessed (IL-1beta, IL-6, IL-10, hs-CRP and TNF-alpha), Pearson correlation will be used to assess the relationship between serum and saliva levels. The investigators will assess whether there is a significant change in the serum levels of endothelial and inflammatory markers and endothelial function using a within-subject paired T-test, with baseline values (low stress) paired with internship stress values (high stress). To assess whether the change in endothelial and inflammatory markers correlate with a change in depressive symptoms, the investigators will utilize a linear regression, with the change in marker level used as explanatory variables and the change in depressive symptoms score (PHQ (change) = mean residency depressive symptoms - baseline depressive symptoms) used as the outcome variable
Examine the temporal relationship between hair cortisol level changes, stress exposure and changes in depressive symptoms | Months 0, 4, 8, 12 of Intern Year
  Statistical analysis will be conducted using Generalized Estimating Equation (GEE) analysis. To assess whether there is a change in hair cortisol indices with internship stress, the investigators will perform a paired T-test, with pre-internship factor cortisol level paired with post-internship factor cortisol level. To determine the relationship between hair-related factors (hair color, hair treatment, washing frequency), transient mediating factors (work hours, outside stressful life events, recent exercise, sleep and illness), long-term mediating factors (BMI, regular exercise schedule, smoking behavior) and long-term cortisol, the investigators will assess whether the difference in level of these factors between the two assessments shows a significant correlation with the difference in cortisol level. Next, the investigators will identify whether that change in hair cortisol is associated with the change in depressive symptoms while accounting for related variables.

CONTACTS AND LOCATIONS:
Overall Officials: Srijan Sen, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Karg K, Sen S. Gene x environment interaction models in psychiatric genetics. Curr Top Behav Neurosci. 2012;12:441-62. doi: 10.1007/7854_2011_184. PMID 22241248
- [Background] Guille C, Sen S. Prescription drug use and self-prescription among training physicians. Arch Intern Med. 2012 Feb 27;172(4):371-2. doi: 10.1001/archinternmed.2011.791. No abstract available. PMID 22371930
- [Background] Guille C, Speller H, Laff R, Epperson CN, Sen S. Utilization and barriers to mental health services among depressed medical interns: a prospective multisite study. J Grad Med Educ. 2010 Jun;2(2):210-4. doi: 10.4300/JGME-D-09-00086.1. PMID 21975622
- [Background] Sen S, Kranzler HR, Krystal JH, Speller H, Chan G, Gelernter J, Guille C. A prospective cohort study investigating factors associated with depression during medical internship. Arch Gen Psychiatry. 2010 Jun;67(6):557-65. doi: 10.1001/archgenpsychiatry.2010.41. Epub 2010 Apr 5. PMID 20368500
- [Background] Karg K, Burmeister M, Shedden K, Sen S. The serotonin transporter promoter variant (5-HTTLPR), stress, and depression meta-analysis revisited: evidence of genetic moderation. Arch Gen Psychiatry. 2011 May;68(5):444-54. doi: 10.1001/archgenpsychiatry.2010.189. Epub 2011 Jan 3. PMID 21199959